CLINICAL TRIAL: NCT01336829
Title: A Phase I, Open Label, Randomized, 2-Panel, 2-Way Crossover Trial to Investigate the Pharmacokinetic Interaction Between Etravirine or TMC278 and Telaprevir at Steady-State in Healthy Subjects.
Brief Title: TMC125IFD1001 - Drug-Drug Interaction of Etravirine With Telaprevir and TMC278 With Telaprevir.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR017989; TMC125IFD1001 (Other: Tibotec Pharmaceuticals, Ireland)
Record Dates: First submitted 2011-04-07; First posted 2011-04-18 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Hepatitis C; HIV
Keywords: Hepatitis C; HIV; TMC125IFD1001; TMC125; Intelence; etravirine; ETR; TMC278; telaprevir; TVR; VX-950; healthy volunteers; crossover
MeSH Terms: conditions — Hepatitis C | interventions — Rilpivirine; telaprevir

ARMS (4):
- 001 (Experimental): ETR/telaprevir Treatment A: ETR 200 mg twice a day from Day 1 to Day 10 + a single dose in the morning on Day 11. Treatment B: telaprevir 750 mg every 8 hours from Day 1 to Day 17 + 2 doses (morning and afternoon) on Day 18 and ETR 200 mg twice a day from Day 8 to Day 17 + a single dose in the morning on Day 18.
  Interventions: Drug: ETR/telaprevir
- 002 (Experimental): telaprevir/ETR Treatment A: ETR 200 mg twice a day from Day 1 to Day 10 + a single dose in the morning on Day 11. Treatment B: telaprevir 750 mg every 8 hours from Day 1 to Day 17 + 2 doses (morning and afternoon) on Day 18 and ETR 200 mg twice a day from Day 8 to Day 17 + a single dose in the morning on Day 18.
  Interventions: Drug: telaprevir/ETR
- 003 (Experimental): TMC278/telaprevir Treatment C: TMC278 25 mg once day from Day 1 to Day 11. Treatment D: telaprevir 750 mg every 8 hours from Day 1 to Day 18 and TMC278 25 mg once daily from Day 8 to Day 18.
  Interventions: Drug: TMC278/telaprevir
- 004 (Experimental): telaprevir/TMC278 Treatment C: TMC278 25 mg once day from Day 1 to Day 11. Treatment D: telaprevir 750 mg every 8 hours from Day 1 to Day 18 and TMC278 25 mg once daily from Day 8 to Day 18.
  Interventions: Drug: telaprevir/TMC278

INTERVENTIONS:
Drug: ETR/telaprevir — Treatment A: ETR 200 mg twice a day from Day 1 to Day 10 + a single dose in the morning on Day 11. Treatment B: telaprevir 750 mg every 8 hours from Day 1 to Day 17 + 2 doses (morning and afternoon) on Day 18, and ETR 200 mg twice a day from Day 8 to Day 17 + a single dose in the morning on Day 18.
  Arms: 001
Drug: TMC278/telaprevir — Treatment C: TMC278 25 mg once day from Day 1 to Day 11. Treatment D: telaprevir 750 mg every 8 hours from Day 1 to Day 18, and TMC278 25 mg once daily from Day 8 to Day 18.
  Arms: 003
Drug: telaprevir/ETR — Treatment A: ETR 200 mg twice a day from Day 1 to Day 10 + a single dose in the morning on Day 11. Treatment B: telaprevir 750 mg every 8 hours from Day 1 to Day 17 + 2 doses (morning and afternoon) on Day 18, and ETR 200 mg twice a day from Day 8 to Day 17 + a single dose in the morning on Day 18.
  Arms: 002
Drug: telaprevir/TMC278 — Treatment C: TMC278 25 mg once day from Day 1 to Day 11. Treatment D: telaprevir 750 mg every 8 hours from Day 1 to Day 18, and TMC278 25 mg once daily from Day 8 to Day 18.
  Arms: 004

SUMMARY:
The purpose of this study is to see the effect of etravirine or TMC278 on how telaprevir is absorbed into the body and the effect of telaprevir on how etravirine or TMC278 are absorbed into the body when administered together.

DETAILED DESCRIPTION:
This is an open-label, randomized, single-dose, crossover trial in healthy volunteers. Crossover means that participants may receive different interventions sequentially during the trial. Randomized means that you will be assigned to a treatment sequence by chance, like flipping a coin. Open-label means that you and your physician will know what treatment you will receive. The study will consist of 3 phases: a screening phase, a treatment phase and a follow-up phase. Total study duration for an individual participant will be approximately 11 weeks. Once found eligible after the screening phase, participants will take part in one of the two parts of the treatment phase. In the first part, a group of 16 participants will receive two treatment sessions, A and B. The order in which the treatments are given will be determined by chance. In treatment A, 200 mg (2 tablets) ETR (etravirine) will be given twice a day from day 1 to 10 with a morning dose only on day 11. In treatment B, 750 mg (2 tablets) TVR (telaprevir) will be given from day 1 to 17 every 8 hours with a morning and afternoon dose only on day 18 and 200 mg ETR will be given twice a day from day 8 to 17 with a morning dose on day 18. In between the 2 sessions, there will be at least 14 days. In the second part, another group of 16 participants will receive 2 treatment sessions, C and D. The order in which these treatments are given will be determined by chance. In treatment C, 25 mg (1 tablet) TMC278 will be given once a day from day 1 to 11. In treatment D, 750 mg (2 tablets) TVR (telaprevir) will be given from day 1 to 18 every 8 hours and 25 mg TMC278 will be given once a day from day 8 to 18. In between the 2 sessions, there will be at least 14 days. All treatments will be taken food. In treatments A and C, participants will come to the unit the day before dosing and in the mornings of day 1, 9 and 10 and for a whole day on day 11. Only in treatment C, overnight stay from day 11 to day 12 is foreseen. In treatment B, participants will come to the unit the day before dosing and in the mornings of days 1, 5, 6, 8, 16 and 17 and for a whole day on days 7 and 18. In treatment D, participants will come to the unit the day before dosing and in the mornings of days 1, 5, 6, 8, 12, 16 and 17 and for a whole day on days 7 and 18 with overnight stay from day 18 to 19. Five to 7 days after last dosing, participants will have a last follow-up visit at the unit (follow-up phase). During the study, safety will be monitored, and during the treatment phase, at specified timepoints, blood samples will be taken for pharmacokinetic evalutions (effect of the body on the drugs). In treatment A, 2 tablets ETR will be given twice a day from day 1 to 10 with a morning dose on day 11. In treatment B, 2 tablets TVR will be given every 8 hours from day 1 to17 with only 2 doses on day 18 and 2 tablets ETR twice a day from day 8 to 17 with a morning dose only on day 18. In treatment C, 1 tablet TMC278 will be given oncy a day from day 1 to 11. In treatment D, 2 tablets of TVR will be given every 8 hours from day 1 to 18 and 1 tablet TMC278 once a day from day 8 to 18.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months prior to selection
* A Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.5 to 30.0 kg/m2
* Healthy on the basis of physical examination, medical history, vital signs, electrocardiogram and clinical laboratory tests performed at Screening
* Women must be postmenopausal for at least 2 years or be surgically sterile or be not heterosexually active for the duration of the study, or have a vasectomized partner, or if of childbearing potential and heterosexually active, be practicing a highly effective method of birth control.

Exclusion Criteria:

* History or evidence of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use, which in the investigator's opinion would compromise the participant's safety and/or compliance with the study procedures
* A positive urine drug test at Screening
* Use of disallowed therapies: concomitant medication, including over-the-counter products, herbal preparations and dietary supplements
* History of significant drug allergy
* Received an investigational drug or used an investigational medical device within 60 days preceding the first intake of study medication or having previously participated in a study with either ETR, TMC278, telaprevir.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Bloodlevels of telaprevir following co-administration with ETR | Over 8 hours on day 18 of treatment B.
Bloodlevels of telaprevir following co-administration with TMC278 | Over 8 hours on day 18 of treatment B.
Bloodlevels of ETR following co-administration with telaprevir | Over 12 hours on day 18 of treatment B.
Bloodlevels of TMC278 following co-administration with telaprevir | Over 24 hours on day 18 of treatment D

SECONDARY OUTCOMES:
Number of participants with adverse events and the severity of adverse events | Over approximately 11 weeks
Bloodlevels of ETR in function of variations of 2 genes (CYP2C9 and CYP2C19) | 1 bloodsample on day 1 of treatment A.
Observed values and changes from baseline for abnormal values of laboratory results. | Over approximately 11 weeks
Observed values and changes from baseline for electrocardiograms (interpretation of electrical activity of the heart) | Over approximately 11 weeks
Evaluation of pulse and blood pressure values, based on changes from baseline and the percentage of participants with values beyond clinically important limits | Over approximately 11 weeks
Physical examination findings and changes from baseline. | Over approximately 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (1):
- Antwerp, Belgium

REFERENCES:
- [Derived] Kakuda TN, Leopold L, Nijs S, Vandevoorde A, Crauwels HM, Bertelsen KM, Stevens M, Witek J, van Delft Y, Tomaka F, Hoetelmans RM. Pharmacokinetic interaction between etravirine or rilpivirine and telaprevir in healthy volunteers: A randomized, two-way crossover trial. J Clin Pharmacol. 2014 May;54(5):563-73. doi: 10.1002/jcph.245. PMID 25975423